CLINICAL TRIAL: NCT07241052
Title: Evaluating Safety and Efficacy of Oral-Spray Bacillus Probiotic (LiveSpo® Smile CARE) in the Prevention and Adjunctive Treatment of Dental Caries in Children
Brief Title: Oral-Spray Bacillus Spore Probiotic in Preventing and Supporting Treatment of Dental Caries in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Collaborators: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TNLS.2025.S
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries
Keywords: Dental caries; Children; probiotics; Oral health; Oral-spray; Bacillus spores
MeSH Terms: conditions — Dental Caries | interventions — Oral Sprays

STUDY DESIGN:
Intervention Model Description: Blinded, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Smile CARE and placebo are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Smile CARE suspension are unrecognizable to investigators, trainers, caregivers, and paticipants due to opaque plastic container. Only the independent statistician is aware of the group codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants allocated to the placebo group will receive a 0.9% NaCl physiological saline spray (20 mL bottle). The spray will be applied directly to carious teeth and adjacent teeth, with a total of six sprays per application, administered twice daily (morning and afternoon), under teacher supervision. All participants will maintain identical daily oral hygiene practices, including the use of fluoride toothpaste and supervised rinsing with 0.2% sodium fluoride mouthwash once per week. The intervention will be continued for a duration of 3 months.
  Interventions: Drug: oral-spray 0.9% NaCl physiological saline solution
- Smile Care (Experimental): Children will receive LiveSpo® Smile CARE, an oral-spray probiotic containing ≥ 1 × 10⁹ CFU/ mL Bacillus subtilis and Bacillus clausii in 20 mL of 0.9% sodium chloride solution. The spray will be administered with the same dosage, frequency, timing, and supervision as the placebo group. The intervention will be continued for a duration of 3 months.
  Interventions: Combination Product: Smile Care

INTERVENTIONS:
Drug: oral-spray 0.9% NaCl physiological saline solution — The oral-spray 0.9% NaCl physiological saline is prepared by extracting 20 mL from a 500 mL polypropylene bottle of 0.9% NaCl intravenous infusion (B. Braun, Germany; product declaration No. VD-32732-19). The solution is contained in an opaque plastic spray bottle identical to that used for the Smile Care.
  Arms: Placebo
Combination Product: Smile Care — LiveSpo® Smile CARE is manufactured as a Class-A medical device (product declaration No. 250002196/PCBA-HN) in compliance with manufacturing standards approved by the Hanoi Department of Health, Ministry of Health. The product is formulated as a 0.9% NaCl physiological saline solution plus Bacillus subtilis ANA48 and Bacillus clausii ANA39 at total concentration of ≥ 1 × 10⁹ CFU/mL (20 billion CFU/20 mL suspension).
  Arms: Smile Care

SUMMARY:
Despite advances in oral health care, cavities remain highly prevalent worldwide, especially among children. Conventional treatment methods focus on removing damaged tooth tissue but fail to completely eliminate or control pathogenic bacteria in the oral cavity, leading to a high risk of caries recurrence in the same or adjacent teeth. Probiotics are a promising biological therapy that can help restore balance in the oral microbiome.

Among probiotics, Bacillus species are unique because they form spores that make them stable under harsh conditions, such as heat and storage. They can also produce enzymes and natural compounds with antibacterial, anti-inflammatory, and protective effects. These features make Bacillus probiotics strong candidates for oral health applications.

This study is designed to evaluate the safety and efficacy of an oral-spray probiotic containing Bacillus subtilis ANA48 and Bacillus clausii ANA39 (LiveSpo® Smile CARE) in preventing and supporting the treatment of tooth decay in children. We hypothesize that this probiotic spray, when used regularly, will be safe and well-tolerated, while effectively reducing harmful bacteria in the mouth, preventing the progression of cavities, and improving overall oral health.

Study Design:

* Sample Size: 130 participants
* Study Location: a primary school in Hanoi, Vietnam Intervention Description: A total of 130 eligible participants will be randomly assigned to two groups (n = 65 per group).

Placebo Group will receive a 0.9% NaCl physiological saline, spray twice daily (morning and afternoon). Each application consists of two sprays at three sites (both dental arches and the front teeth), for a total of six sprays per use, continued for three consecutive months.

Smile Care Group will receive an oral-spray probiotics containing ≥ 1 billion CFU/mL × 20 mL of Bacillus subtilis and Bacillus clausii (LiveSpo Smile CARE). The dosage, frequency, and duration of use will be the same as in the placebo group.

All participants will receive the same standard dental care throughout the study, including the use of identical toothpaste, supervised weekly fluoride rinsing with 0.2% sodium fluoride (NaF), and scheduled follow-up visits. The probiotic and placebo sprays will be packaged in blinded bottles and administered according to the study protocol to maintain objectivity.

Study Duration: 12-18 months

DETAILED DESCRIPTION:
Tooth decay is one of the most common oral health problems in children. It not only causes pain and discomfort but also interferes with eating, daily activities, and overall quality of life. In severe cases, untreated cavities may progress to pulp infection requiring more complex treatment. One of the major causes of dental caries is an imbalance of the oral microbiome, with Streptococcus mutans being the main pathogen. Improving the oral microbiome provides a safe, long-term strategy for managing cavities, particularly in children, while avoiding the risks of antibiotic resistance.

Bacillus probiotics have been extensively studied for their benefits on gastrointestinal and respiratory health but remain underexplored in the context of oral health. This trial is among the first to evaluate the safety and potential synergistic effects of Bacillus subtilis and Bacillus clausii in improving clinical symptoms, reducing pathogenic bacterial load, and preventing the progression of dental caries after 1, 2, and 3 months of intervention.

This is a randomized, double-blind, placebo-controlled clinical trial conducted over 3 months. A total of 130 primary school children aged 7-10 years (grades 2-4) with diagnosed dental caries will be enrolled. Children will be stratified by age group (7-<8, 8-<9, 9-10 years) and number of decayed teeth (≤2 or >2), then randomized in a 1:1 ratio to receive either: Placebo group and Smile Care group.

Both sprays will be administered twice daily (morning and afternoon), two sprays per site (both dental arches and front teeth), totaling six sprays per use, for three consecutive months.

- Primary Outcome: Changes in clinical symptoms, including Decayed Teeth index using ICDAS classification, Progressive caries rate, Early caries rate and Early caries rate code 1) at months 1 and 3 vs. day 0.

- Secondary Outcomes:

Changes in cytokine levels (ELISA) and semi-quantification of bacterial pathogens (real-time PCR) at months 1 and 3 compared with day 0.

- Exploratory Outcomes: Detection of B. subtilis ANA48 and B. clausii ANA39 in soft dentin and saliva samples (months 1, 2, and 3) of the Smile Care group, but not in the Placebo group.

Comparative analysis of oral microbiota diversity and bacterial density at month 1 between the placebo and Smile Care groups, using a reference group of at least 10 healthy children without dental caries.

Statistical Analysis:

Categorical variables will be analyzed using chi-square or Fisher's exact tests, while continuous variables will be assessed using t-tests, Mann-Whitney U, or Wilcoxon signed-rank tests depending on distribution.

ELIGIBILITY:
Inclusion Criteria:

* Children (male or female) aged 7-10 years, currently enrolled in primary school (grades 2-4).
* At least one decayed tooth (any stage) at the time of screening.
* Commitment to comply with study requirements, including refraining from using any other probiotic products for the ear, nose, and throat that could affect study outcomes.
* Written informed consent obtained from a parent or legal guardian.

Exclusion Criteria:

Participant-level exclusion:

* Presence of severe chronic disease, allergy, or use of antibiotics within 1 month prior to study initiation.
* Use of oral or throat probiotic sprays/lozenges within the past 30 days (excluding gastrointestinal probiotics).
* Participation in another clinical study within the past 30 days.
* Acute oral conditions (e.g., abscess, severe gingivitis) interfering with examination or intervention.
* Currently receiving dental treatment at specialized dental/oral health facilities.
* History of congenital immunodeficiency or infectious disease.
* Psychiatric disorders or sleep disturbances.
* Known sensitivity or allergy to components of the investigational product.

Tooth-level exclusion:

* Hard tissue lesions not caused by dental caries.
* Supernumerary teeth or teeth not part of the functional dental arch.
* Carious teeth with pain lasting >10 seconds during examination.
* Carious teeth with visible pulp hyperemia (high risk of pulp complications).
* Teeth showing signs of pulp disease, pulp necrosis, or periapical pathology.
* Teeth previously treated with endodontic therapy or permanently restored with crowns.
* Primary teeth with mobility grade ≥2 (due to disease or natural exfoliation).

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Decayed Teeth Index | Day 0, and months 1, 2, 3
  Changes will be calculated for each participant based on the following parameters: the number of decayed teeth assessed using the International Caries Detection and Assessment System (ICDAS, codes 0-6), progressive caries rate, early caries rate, and early caries rate (code 1). These parameters will be evaluated at month 3 compared with day 0. Month 1 and Month 2 will be collected as supplementary exploratory timepoints.

SECONDARY OUTCOMES:
Changes in the concentration of pathogenic bacteria in deep carious dentin and saliva samples | Day 0 and months 1, 2, 3
  The semi-quantitative assessment of changes in pathogenic bacteria concentrations (S. mutans, P. gingivalis, and A. actinomycetemcomitans) at month 3 compared with day 0, supplementary timepoints (month 1,2).
Changes in Inflammatory Cytokines and IgA levels in deep carious dentin and saliva samples | Day 0 and months 1, 2, 3
  Measurement of pro-inflammatory cytokine (IL-1β, IL-5, IL-6, IL-8, IL-17, TNF-α or IFN-γ) and IgA concentrations at day 0 and month 3, supplementary timepoints (month 1,2).

OTHER OUTCOMES:
Changes in the oral microbiome at month 1 compared to day 0 | Day 0 and 1 month
  Analysis of the diversity and taxonomy compositions (16S rRNA NGS) of deep carious dentin and saliva samples
Detection of Probiotic Bacillus Spores | Day 0 and months 1, 2, 3
  Detection of Bacillus subtilis and Bacillus clausii spores in the deep carious dentin and saliva at months 1, 2, and 3 using real-time PCR, based on cycle threshold (Ct) values for qualitative assessment of presence.

CONTACTS AND LOCATIONS:
Overall Officials: Nga TT Pham, PhD. MD, Study Chair — Hanoi Medical University; Thu TH Nguyen, Assoc. Prof., Principal Investigator — Hanoi Medical University; Anh TV Nguyen, Assoc. Prof., Principal Investigator — Spobio Research Center, Anabio R&D

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), and clinical study reports (CSR). For more information or to submit a request, please contact anabio.rd2021@gmail.com

REFERENCES:
- [Result] Kim H, Han CY, Eun SH, Kim MG, Im AR, Lee B. Inhibitory effects of Bacillus velezensis ID-A01 supernatant against Streptococcus mutans. BMC Microbiol. 2023 Nov 24;23(1):362. doi: 10.1186/s12866-023-03114-2. PMID 37996837
- [Result] Jindal G, Pandey RK, Agarwal J, Singh M. A comparative evaluation of probiotics on salivary mutans streptococci counts in Indian children. Eur Arch Paediatr Dent. 2011 Aug;12(4):211-5. doi: 10.1007/BF03262809. PMID 21806906
- [Result] Aleti G, Sessitsch A, Brader G. Genome mining: Prediction of lipopeptides and polyketides from Bacillus and related Firmicutes. Comput Struct Biotechnol J. 2015 Mar 24;13:192-203. doi: 10.1016/j.csbj.2015.03.003. eCollection 2015. PMID 25893081
- [Result] Weisser K, Ganz R, Olafsson A, Wyler F, Rutishauser M. Bronchopulmonary dysplasia in the premature baby. Respiration. 1970;27:Suppl:36-40. No abstract available. PMID 4929038
- [Result] Bustamante M, Oomah BD, Mosi-Roa Y, Rubilar M, Burgos-Diaz C. Probiotics as an Adjunct Therapy for the Treatment of Halitosis, Dental Caries and Periodontitis. Probiotics Antimicrob Proteins. 2020 Jun;12(2):325-334. doi: 10.1007/s12602-019-9521-4. PMID 30729452
- [Result] Simon-Soro A, Mira A. Solving the etiology of dental caries. Trends Microbiol. 2015 Feb;23(2):76-82. doi: 10.1016/j.tim.2014.10.010. Epub 2014 Nov 27. PMID 25435135
- [Result] Lu Y, Lin Y, Li M, He J. Roles of Streptococcus mutans-Candida albicans interaction in early childhood caries: a literature review. Front Cell Infect Microbiol. 2023 May 16;13:1151532. doi: 10.3389/fcimb.2023.1151532. eCollection 2023. PMID 37260705
- [Result] Takahashi N, Nyvad B. The role of bacteria in the caries process: ecological perspectives. J Dent Res. 2011 Mar;90(3):294-303. doi: 10.1177/0022034510379602. Epub 2010 Oct 5. PMID 20924061
- [Result] Sampaio-Maia B, Caldas IM, Pereira ML, Perez-Mongiovi D, Araujo R. The Oral Microbiome in Health and Its Implication in Oral and Systemic Diseases. Adv Appl Microbiol. 2016;97:171-210. doi: 10.1016/bs.aambs.2016.08.002. Epub 2016 Sep 21. PMID 27926431